CLINICAL TRIAL: NCT06362096
Title: ve Study of Diarrhea Tolerance of Pyrotinib Combined With Trastumab and Taxane in the First-line Treatment of HER2-positive Advanced Breast Cancer
Brief Title: A Multicenter, Prospective Study of Diarrhea Tolerance of Pyrotinib Combined With Trastumab and Taxane in the First-line Treatment of HER2-positive Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huihua Xiong (Other)
Responsible Party: Sponsor-Investigator, Huihua Xiong, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: pyrotinib diarrhra
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM1 (Experimental)
  Interventions: Drug: Trastuzumab+pyrotinib+taxene

INTERVENTIONS:
Drug: Trastuzumab+pyrotinib+taxene — Trastuzumab (first cycle 8mg/Kg, subsequent 6mg/Kg, iv, q3w) Pyrrotinib * po, qd, q3w The first cycle 240mg+ montmorillonite powder, the second cycle 320mg+ montmorillonite powder prevention Subsequent cycle 400mg+* montmorillonite powder used when necessary taxenes

SUMMARY:
To explore a reasonable and effective way to reduce the incidence of grade 3 or above diarrhea caused by pyrotinib

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years, ≤75 years
2. Her2-positive recurrent or metastatic breast cancer; Patients with local recurrence need to be confirmed by the investigator that radical surgical resection is not possible.
3. Did not receive any systemic antitumor therapy in the advanced stage;
4. At least one measurable lesion was present according to RECIST1.1 criteria.
5. The ECOG score is 0 to 1
6. The functional major organs must be normal
7. Volunteer to participate in this study, sign informed consent, have good compliance and willing to cooperate with follow-up

Exclusion Criteria:

1. Have received any systematic antitumor therapy at the recurrence/metastasis stage;
2. Tyrosine kinase inhibitor (TKI) formulations targeting HER have been used at any stage of breast cancer
3. Patients judged by the investigators to be unsuitable for systematic chemotherapy.
4. Patients with active brain metastases (meaning those requiring mannitol treatment or with symptomatic brain metastases);
5. Had undergone major surgical procedures or significant trauma within 4 weeks prior to randomization, or were expected to undergo major surgical treatment.
6. Serious heart disease or discomfort
7. Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors that affect the use and absorption of medications.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of ≥ grade 3 diarrhea | Up to 2 years
  Incidence of ≥ grade 3 diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Xiong huihua, Principal Investigator — Tongji Hospital Affiliated of Tongji Medical College Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided